CLINICAL TRIAL: NCT04705987
Title: Randomized Double-blind Trial to Study the Benefit of Colchicine in Patients With Acutely Decompensated Heart Failure
Acronym: COLICA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMIB-CO-2020-01
Record Dates: First submitted 2021-01-11; First posted 2021-01-12 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-09

CONDITIONS: HEART FAILURE
MeSH Terms: conditions — Heart Failure | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Colchicine 0.5 mg
  Interventions: Drug: Colchicine 0.5 MG
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 MG — Colchicine 0.5 mg/24h Treatment 8 weeks
  Arms: Experimental
Drug: Placebo — Placebo 1c/24h Treatment 8 weeks
  Arms: Placebo

SUMMARY:
Heart failure (HF) is a chronic disease associated with multiple acute decompensations, which are the main cause of hospital admission above 65 years and two thirds of the high costs associated with the disease. Furthermore, in the patient they reflect a phase of clinical instability, with a higher risk of early readmission (20-30% at 30 days) and higher mortality (10-15% at 30 days and 30-40% at 1year).

However, the investigators do not have treatments specifically aimed at this unstable phase, known as acute or decompensated (HF). It is known that, in this acute and unstable state, there is an increase in inflammatory parameters. Indeed, our group has recently demonstrated the relevance of the interleukin-1 axis, in particular IL-1beta and sST2 concentrations identified a worse prognosis regardless of HF phenotype. Colchicine, a widely available drug, has proven to be a powerful cardiovascular anti-inflammatory, acting on inflammasome and therefore inhibiting the production of IL1-beta.The study hypothesis is that colchicine administered early during the acute phase can promote stability in terms of biomarkers of cardiac function and new decompensations. For this it is designed a randomized, double-blind clinical study with two arms (colchicine 0.5 mg vs. placebo) initiated within the first 24 hours of hospitalisation and administered for 60 days, in patients with acute decompensated HF with either reduced or preserved LV ejection fraction.

DETAILED DESCRIPTION:
The primary objective of the study is the reduction of NT-proBNP at two months of treatment. A secondary objective is to attain a greater clinical stability, in terms of reduction of new HF decompensations and need for diuretics, and symptoms improvement. The calculated population size is 278 patients. Follow-up visits will be carried out at discharge, 7 days, 4 weeks and 8 weeks after the hospital discharge. The potential of the study is very high given the high prevalence and clinical impact of HF hospitalizations, together with the absence of specific treatment for this phase of the disease. Therefore, in case of a positive result, this would mean a huge clinical, social and health benefits, as well as being an important therapeutic progress.

ELIGIBILITY:
Inclusion Criteria:

1. Unscheduled visit for symptoms and / or congestive signs of HF that require treatment with intravenous diuretics (at least 40 mg intravenous furosemide)
2. Clinical evidence, by symptoms or signs, and / or radiological of congestion.
3. NT-proBNP concentration greater than 900 pg / ml at screening visit.
4. Age over 18 years.
5. Patients who have given their informed consent in writing.

Exclusion Criteria:

1. Severe valve disease with indication for surgical repair.
2. Extracardiac disease with estimated vital prognosis of less than 1 year.
3. Inflammatory bowel disease (Crohn's disease or ulcerative colitis), diarrhea chronic or malabsorption.
4. Rheumatic inflammatory disease.
5. Serious gastrointestinal disorders
6. Stomach ulcer
7. Hematological disorders, such as blood dyscrasias
8. Previous neuromuscular disease
9. Severe renal failure (glomerular filtration rate <30 ml / kg / min / 1.73m2)
10. History of cirrhosis, chronic active hepatitis or severe liver disease, defined by GOT (AST) or GPT (ALT) values that exceed 3 x upper limit of normality
11. Patient who is taking colchicine for other indications (mainly chronic prescriptions for familial Mediterranean fever or gout). No washout period will be required for patients who have been treated with colchicine and have stopped treatment prior to randomization.
12. Patient with a history of allergic reactions or significant sensitivity to colchicine.
13. Chronic treatment with immunosuppressants, corticosteroids, interleukin-1 antagonists in the 6 months prior to inclusion.
14. Pregnant or lactating women, where pregnancy is defined as the state of a woman after conception and until the end of gestation, confirmed by a positive test result for human chorionic gonadotropin (hCG), or planned become pregnant or plan to breastfeed during study treatment or within 30 days of the end of study drug treatment.
15. Woman of childbearing potential who is unwilling to inform her partner of her participation in this clinical study or to use 2 effective contraceptive methods that are acceptable or to practice strict sexual abstinence (the investigator must assess the reliability of sexual abstinence and make it the preferred and usual lifestyle of the subject) during treatment with study drug (colchicine or placebo) and for an additional 30 days after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Decreased NT-proBNP levels | Up to 8 weeks
  Decreased (N-terminal prohormone of brain natriuretic peptide) levels

SECONDARY OUTCOMES:
Improvement of clinical stability | Up to 8 weeks
  dose of intravenous diuretics
Improvement of clinical stability | Up to 8 weeks
  NYHA (New York Heart Association) Scale . Level 1 to 4. Level 1 is the one with the least limitation or symptoms.
Improvement of clinical stability | Up to 8 weeks
  EVA scale . Level 1 to 10 . Level 1 is the one with the least pain, limitation or symptoms.
Improvement of clinical stability | Up to 8 weeks
  LIKERT scale. Level 1 to 5 . Level 1 expresses the patient's agreement with a specific aspect.
Improvement of clinical stability | Up to 8 weeks
  Number of Acute Decompensation Episodes
Improvement of clinical stability | Up to 8 weeks
  Number of Congestion Episodes
Improvement of clinical stability | Up to 8 weeks
  biomarkers (hsTnT, IL-1 beta, IL-6, sST2 y CA125.)
Mortality rate reduction | Up to 8 weeks
Total days of hospitalization | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Domingo Pascual Figal, MD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Spain